CLINICAL TRIAL: NCT06291935
Title: A Prospective, Open-label, Phase 1b, Single-arm, Safety Study of an Intravitreal Application of a Recombinant Adeno-associated Virus Vector Expressing CNGA1 (AAV2.NN-CNGA1) in Patients With Retinitis Pigmentosa Due to CNGA1 Mutations
Brief Title: Safety and Tolerability of Intravitreal Administration of VG901 in Patients With Retinitis Pigmentosa Due to Mutations in the CNGA1 Gene
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: VeonGen Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VG901-2021 A; EU CT: 2023-504383-42-00 (Other: EMA)
Record Dates: First submitted 2024-02-01; First posted 2024-03-04 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Retinitis Pigmentosa
Keywords: CNGA1 mutation; AAV2; Gene Therapy; Eye disease
MeSH Terms: conditions — Retinitis Pigmentosa; Eye Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- VG901 (Experimental): Participants will receive a single dose of intravitreal injection of VG901 in most affected eye at Day 0.
  Interventions: Drug: VG901

INTERVENTIONS:
Drug: VG901 — Administered as specified in the treatment arm. Study Cohort 1 - Low dose; Study Cohort 2 - High dose
  Other Names:
  Gene Therapy (AAV2.NN-CNGA1)
  Other Names: AAV2.NN-CNGA1

SUMMARY:
The goal of this phase 1 clinical trial is to learn about the safety and efficacy of a gene therapy, VG901, in patients with a rare disorder of the eye called Retinitis Pigmentosa. The main questions the study aims to answer are:

* What is the best tolerated dose and are there any side effects, in particular any inflammatory reactions post drug administration?
* Are there any early signs of efficacy on visual function?

Participants will be administered a single intravitreal dose of VG901 into the most affected eye through a syringe and followed up for a year to monitor safety and efficacy. There will be two cohorts of participants in this study. Study Cohort 1 will receive the low dose and Study Cohort 2 will receive the high dose as specified in the Protocol.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for study entry, subjects must satisfy all the following criteria:

1. Able to understand and willing to consent to study participation by a written informed consent
2. Male or female ≥ 18 years of age
3. Clinical diagnosis of RP
4. Confirmed pathogenic, biallelic variants in the CNGA1 gene
5. Ellipsoid zone (EZ) length of the fovea of ≥ 3000 μm in the study eye

Exclusion Criteria:

Subjects will be excluded from the study if one or more of the following statements are applicable to either eye:

1. Additional interfering ocular conditions which would impact study results (e.g., ocular opacity and advanced cataract, uveitis, amblyopia)
2. History or presence of glaucoma
3. Ocular surgery, intravitreal or subretinal implantation of a medical device (within 6 months of screening)
4. Mutations known to cause inherited retinal disease other than biallelic variants in the CNGA1 gene
5. History of ocular infection with herpes simplex virus
6. History of ocular malignancies
7. History of disorders of the internal retina (e.g., retinal detachment)
8. Patients with uncontrolled diabetes (HbA1c > 7%)
9. Any other retinopathy due to other diseases - including, but not limited to arterial hypertension, previous vascular retinal occlusion, trauma or acquired inflammatory diseases, contraindication to pharmacological mydriasis (e.g., history of angle block glaucoma), diabetes (diabetic retinopathy including macular oedema)
10. Absence of visual function on the contralateral eye
11. Any damage to the optic nerve
12. Individuals performing any other therapy for RP within 3 months before the study, such as - but not limited to - transcorneal electrostimulation
13. Systemic conditions (e.g., autoimmune disorders) which may affect study participation or outcome measures
14. History of immunodeficiency or other medical conditions which may increase the risk of VG901 administration
15. Systemic illness (e.g., hepatitis or human immunodeficiency virus [HIV] infection) or medically relevant abnormal laboratory values (3 x upper limit of normal [ULN]) in blood analysis including renal and hepatic function
16. Current, or recent, participation in other study/ or administration of investigational biologic agent within 3 months of Screening; Use of any investigational agent, or systemic corticosteroids, or other immunosuppressive drug(s) within 3 months before Screening
17. History of allergy or sensitivity to any compound used in the study
18. Contraindications to systemic immunosuppression
19. Subjects with increased risk of bleeding (i.e., use of anticoagulants or anti-platelet agents within 7 days before VG901 administration and subjects with international normalized ratio > 2 or Quick < 50% or partial thromboplastin time > 50 seconds, thrombocytopenia, as well as any other known coagulopathy)
20. Subject/partner of childbearing potential unwilling to use adequate contraception for the period between Screening and 30 days after treatment, defined as the period from Screening until 30 days after treatment (defined as administration of therapeutic to the eye)
21. For females of childbearing potential, a positive pregnancy test at Screening or Baseline
22. Females who are breastfeeding
23. Previous receipt of any AAV gene therapy product
24. Any condition which leads the investigator to believe that subject cannot comply with the protocol requirements or that may place the subject at an unacceptable risk from participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline to Month 12
  Number of Adverse Events (AEs) and Serious Adverse Events (SAEs). Ocular inflammation is defined as an adverse event of special interest (AESI). AESI follow the same reporting requirements as SAE.

SECONDARY OUTCOMES:
Physical Examination | Screening to Month 12
  A complete physical examination will be done at Screening and at Baseline and then at Month 12. On the other timepoints during the 1-year active follow-up phase, symptom-directed physical examination will be conducted. Abnormal examination results will be recorded.
Pulse rate | Screening to Month 12
  Will be recorded in beats per minute.
Blood pressure | Screening to Month 12
  Systolic and diastolic blood pressure will be recorded in mmHg.
Body temperature | Screening to Month 12
  Will be recorded in °C.
Respiratory rate | Screening to Month 12
  Will be recorded in breaths per minute.
Slit lamp examination | Screening to Month 12
  Abnormal examination results of conjunctiva, cornea, sclera, lens, anterior segment, and anterior chamber cells as well as quantification of vitreous inflammation and grading of anterior chamber flare will be recorded.
Fundus biomicroscopy | Screening to Month 12
  Cup-to-Disc (C/D) ratio and abnormal examination results will be recorded.
Optical coherence tomography (OCT) | Screening to Month 12
  Abnormal examination results will be recorded.
Fundus autofluorescence | Screening to Month 12
  Abnormal examination results will be recorded.
Tonometry | Screening to Month 12
  Intraocular Pressure (IOP) will be recorded in mmHg.
Adeno-associated virus (AAV) spread | From Baseline until two consecutive samples test negative
  As detected by quantitative polymerase chain reaction (qPCR) in peripheral blood, urine, and tear. Recorded in vector copies per µL of fluid DNA.
Immunopathology | Baseline to Month 12
  Using specific enzyme-linked immunosorbent assays (ELISA) for humoral antibodies against rAAV2 capsid protein.

CONTACTS AND LOCATIONS:
Overall Officials: Katarina Stingl, Principal Investigator — Center for Ophthalmology, University of Tuebingen
Locations (1):
- Center for Ophthalmology, University of Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No